CLINICAL TRIAL: NCT05682118
Title: Impact of Dynamic CoROnary RoADmap System for Guidance of Instantaneous Wave-Free Ratio or Fractional Flow Reserve: A Single-Center, Randomized Study (ROAD-IFR Trial)
Brief Title: Impact of Dynamic CoROnary RoADmap System for Guidance of Instantaneous Wave-Free Ratio or Fractional Flow Reserve
Acronym: ROAD-IFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Yongcheol Kim, Clinical Associate Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9-2022-0134
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Heart Disease
Keywords: iFR/FFR; Roadmap
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: The sample size was calculated using effect size (Cohen's d) for the effectiveness of the dynamic coronary roadmap system for the guidance of the iFR and FFR. The effect size was assumed to be 0.4, which is a small to medium effect size. The sample size of 113 participants for each group was estimated to provide 90% power with a 2-sided type I error of 0.05.
  This is a single-center randomized study and will be conducted in 226 patients with 50-90% coronary artery stenosis on angiography. Afterward, randomly assigned, 113 patients will be tested using the roadmap system, and 113 patients will be tested without using the roadmap system. Methods for measuring FFR and iFR and all PCI will use standardized testing and procedure methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tested using the roadmap system (Experimental): tested using the roadmap system
  Interventions: Procedure: roadmap; Procedure: iFR/FFR
- tested without using the roadmap system (Active Comparator): tested without using the roadmap system.
  Interventions: Procedure: iFR/FFR

INTERVENTIONS:
Procedure: roadmap — FFR and iFR tests using the roadmap system, or FFR and iFR tests without using the roadmap system.
  Pressure wire into guiding catheter The equalization of the pressure wire with the aortic pressure(after placing the pressure wire on the tip of the guiding catheter and removal of contrast media by saline flushing) and the placement of the pressure wire on the distal of the blood vessel to measure iFR. After iFR measurement, the pressure wire was pulled back into the tip of the guiding catheter to check the presence of pressure drift. A final Pd/Pa between 0.97 and 1.03 is considered acceptable. Following confirming no pressure drift, a mode change will be done from iFR to FFR, and then a re-check of the time between the equalization of the pressure wire with the aortic pressure will be planned. In all lesions, FFR value were measured with hyperemia, achieved by intracoronary (IC) bolus injection of nicorandil (Sigmart®; Chugai Pharmaceutical Co., Ltd., Tokyo, Japan) 2 mg.
  Arms: tested using the roadmap system
Procedure: iFR/FFR — Patients undergoing pressure wire test with moderate stenosis. Pressure wire into guiding catheter The equalization of the pressure wire with the aortic pressure(after placing the pressure wire on the tip of the guiding catheter and removal of contrast media by saline flushing) and the placement of the pressure wire on the distal of the blood vessel to measure iFR. After iFR measurement, the pressure wire was pulled back into the tip of the guiding catheter to check the presence of pressure drift. A final Pd/Pa between 0.97 and 1.03 is considered acceptable. Following confirming no pressure drift, a mode change will be done from iFR to FFR, and then a re-check of the time between the equalization of the pressure wire with the aortic pressure will be planned. In all lesions, FFR value were measured with hyperemia, achieved by intracoronary (IC) bolus injection of nicorandil (Sigmart®; Chugai Pharmaceutical Co., Ltd., Tokyo, Japan) 2 mg.

SUMMARY:
In patients with 50-90% stenosis of the coronary artery, the coronary roadmap (dynamic roadmap) is performed when the conventional fractional flow reserve (FFR) and instantaneous wave-free ratio (iFR) are performed. coronary roadmap system) to confirm the effectiveness of the function.

DETAILED DESCRIPTION:
In coronary angiography, 50% or more stenosis of the causative vessel is observed in a patient with stable angina pectoris (SAP) or 50% or more stenosis of a non-causative vessel is observed in acute coronary syndrome (ACS) Based on 0.90, if it is less than 0.89, PCI is performed, and if it is 0.90 or more, drug treatment is performed. When the pressure wire tests are performed, the pressure wire is inserted from the origin of the blood vessel through the lesion to the distal portion, and the pressure wire is placed at the distal end of the blood vessel for measurement. In this process, there are many cases where the pressure wire escapes the branch blood vessel or does not pass through well. It takes a long time to stand up and evaluate stenosis, and in many cases, an additional contrast medium is used to additionally check blood vessel travel and to check the position and condition of the pressure wire. To overcome this, the software roadmap installed in the cardiac fluoroscopy device of the cardiac catheterization room can be helpful. However, there are currently no studies related to roadmaps in coronary artery examination. Therefore, in this study, we want to evaluate the effectiveness of the roadmap when examining FFR and iFR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years or older
2. Patients with stable angina, including asymptomatic ischemic heart disease, who have 50-90% stenosis of the causative vessel by coronary angiography
3. Acute coronary syndrome patients with multivessel disease and 50-90% stenosis of non-caused vessels that did not cause acute coronary syndrome
4. Patients who voluntarily decided to participate in this study and gave written consent to the subject consent form

Exclusion Criteria:

1. Patients with acute coronary syndrome and single vessel disease
2. Patients who have undergone previous coronary artery bypass grafting
3. Poor coronary blood flow (TIMI grade ≤ 2)
4. If life expectancy is less than one year
5. Women who are pregnant or wish to become pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
iFR time | Through procedure completion, up to 24 hours
  iFR time: the time interval between the pressure wire into the guiding catheter and the placement of the pressure wire on the distal of the blood vessel to measure iFR
FFR time | Through procedure completion, up to 24 hours
  FFR time: the time interval between the equalization of the pressure wire for FFR and the placement of the pressure wire on the distal of the blood vessel to measure FFR

SECONDARY OUTCOMES:
Success rate of placement of the pressure wire on the distal of the blood vessel to measure iFR/FFR | Through procedure completion, up to 24 hours
  The success rate of advancing pressure wire to a target vessel distally
Use of contrast medium until the pressure wire is advanced to the distal end of the blood vessel | Through procedure completion, up to 24 hours
  Use of contrast medium until the pressure wire is advanced to the distal end of the blood vessel
The amount of contrast medium used until the pressure wire is advanced to the distal end of the blood vessel | Through procedure completion, up to 24 hours
  The amount of contrast medium used until the pressure wire is advanced to the distal end of the blood vessel
Total procedure time to assess functional significance using iFR/FFR pressure wire | Through procedure completion, up to 24 hours
  Total procedure time between insertion and out of guiding catheter via a sheath
Total procedure time | Through procedure completion, up to 24 hours
  Total procedure time
Total amount of contrast media usage | Through procedure completion, up to 24 hours
  Total amount of contrast media usage
Total dose of radiation exposure | Through procedure completion, up to 24 hours
  Total dose of radiation exposure
Complications related to the procedure | Through procedure completion, up to 24 hours
  Complications related to the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yongcheol Kim, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
The data set is available from the the corresponding author upon reasonable request.